CLINICAL TRIAL: NCT02082002
Title: Multidimensional Assessment of Fatigue in Multiple Sclerosis- Observational Study - Ticino
Status: Completed | Type: Observational
Sponsor: Claudio Gobbi (Other Government)
Collaborators: Swiss Multiple Sclerosis Society (Unknown)
Responsible Party: Sponsor-Investigator, Claudio Gobbi, Dr med., Vice head physician, Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Other Study IDs: EOC.NSI.13.02
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple scerlosis; Fatigue; Sleep; Somnolence; Depression; Cognitive disorders
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleepiness; Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MS-Group: MS-Group
- Healthy control: Healthy control

SUMMARY:
Fatigue is a common symptom in patients with multiple sclerosis, however, its nature is not completely understood. Fatigue overlaps often with other symptoms such as somnolence, depression and cognitive disorders, from which it is not always readily distinguished. The evaluation of fatigue and the three most frequently associated symptoms using a multidimensional approach might allow to understand, which methodology is the best indicated to estimate the prevalence of fatigue with greatest accuracy, leading to a better differentiation of the symptoms in the diagnostic setting.

DETAILED DESCRIPTION:
Objectives: 1- to provide a detailed characterization of fatigue in a cohort of selected MS patients, including a definition of the boundaries and the overlaps between fatigue, somnolence, mood disorders and attention dysfunction; 2- to see how the prevalence and the overlaps between fatigue, somnolence, depression and attention dysfunction are influenced by the method of assessment. 3-To better characterize the sleep structure in MS patients with fatigue under both the macro- and microstructural point of view.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of MS (14,15) or CIS (16);according to the most recent standard criteria
* Expanded Disability Status Scale (EDSS) score < 7.0 (17);
* Last magnetic resonance imaging (MRI) within the previous 12 months;
* Male or female;
* >18 years old;
* Willing to perform the study procedures;
* Signed Informed consent.

Exclusion Criteria:

* Mini Mental Status Examination (MMSE) score < 24;
* Relapse within the last 3 months;
* Radiologically isolated syndrome (RIS);
* History of drug and/or alcohol abuse;
* Any serious general medical condition like decompensated cardiopulmonary disease, cancer or decompensated renal failure, as well as any neurological condition (other than MS) that can interfere with the correct execution of the study design.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 1 Day
  a self-administered 9-items scale. The patient gives a score from 1 to 7 to each item. The resulting score is given as the mean value. Subjects with a score higher that 4 are considered fatigued. This scale assesses the impact of fatigue on multiple outcomes, with a physical focus. FSS has been validated for MS, it has an acceptable internal consistency, it is a reliable, completely safe and brief scale, which in addition has been shown to follow clinical changes in fatigue perception over time. Furthermore, FSS scores correlate with other commonly used fatigue scales, like the Modified Fatigue Impact Scale

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale | 1 Day
  a 21-items scale, which was proposed by the MS Council for Clinical Practice Guidelines as a shortened version of the previous 40-items Fatigue Impact Scale (21). The patient gives a score from 0 to 4 at each item, to express how every item best describes the personal experience, where 0 is "never" and 4 is "almost always"; the final score is the sum of the 21 items. The cut-off score beyond whom the subject can be considered fatigued is 38. The administration time is approximately 5-10 minutes. The MFIS is a structured, reliable, self-report questionnaire that the patient can generally complete easily, with little or no intervention from an interviewer. It provides a multidimensional assessment of fatigue, considering its impact on physical (9 items), cognitive (10 items) and phychosocial (2 items) functioning in daily life. It has a good reproducibility and a strong correlation with FSS results
Fatigue Scale for Motor and Cognitive functions | 1 Day
  a validated questionnaire specifically developed for MS (22). It is a 20-items scales that allows graduation of fatigue severity, and separate evaluation of motor (10 items) and cognitive (10 items) fatigue components. The response pattern for each item consists in a five-point Likert scale; a total score higher than 43 indicates the presence of mild fatigue and the score increases proportionally to the severity of fatigue (> 53: moderate; >63 severe); the cut-off for both the cognitive and the motor subscales is 22. FSMC provides good reliability and correlates with both FSS and MFIS scores
Visual analogue scale for fatigue | 1 Day
  a simple and quick measure of the patient's instant perception of fatigue on him/herself. It is a measurement of the impression at the moment of the interview. It consists of a graphic 10 cm wide line with "no fatigue" at one end and "very severe fatigue" on the other and the subject is asked to place a cross at the point that best express his/her answer to the question "how do you feel in this moment?"
Maintenance of wakefulness test | 1 Day
  it objectively explores somnolence in terms of ability to remain awake in sleep- promoting environmental conditions. It has to be performed after a nocturnal PSG recording because the knowledge of the previous sleep is essential for MWT interpretation. Recordings include only EEG, EMG and EOG from the previous PSG and are carried out in a dim room, with slight illumination. Patients are instructed to stay awake as long as possible. Four sessions are recorded every two hours, each lasting until the patient falls asleep or for 40 minutes of continuous awake state. The sleep latency is assessed in each of the four recordings and it is defined by the elapse time in minutes on each trial before sleep onset: the patient is considered asleep after three 30 seconds EEG epochs of stage N1 of non-REM sleep, or one 30-second epoch of any other sleep stage.
Epworth Sleepiness Scale | 1 Day
  a self-administered questionnaire with 8 questions, which provide a measure of a subject's general level of daytime sleepiness (26). Subjects are required to indicate their chance to fall asleep in 8 different situations on a rating scale from 0 to 3, where 0 means no chance and 3 big chance. The total score is the sum of the eight items, and a score higher that 10 suggests an excessive daytime sleepiness, whose severity increases proportionally to the score. Most people can answer the questions with no assistance in less than 5 minutes.
Visual analogue scale for somnolence | 1 Day
  a simple and quick measure of the patient's instant perception of somnolence on him/herself. It is a measurement of the impression at the moment of the interview. It consists of a graphic 10 cm wide line with "no sleepiness" at one end and "very severe sleepiness" on the other and the subject is asked to place a cross at the point that best express his/her answer to the question "how do you feel in this moment?".
Beck depression inventory II | 1 Day
  a 21-item self-report of depressive symptomatology for individuals aged 13 to 80 years (32). It was developed to have clinical sensitivity for assessing depression criteria reported in the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV) and intends to assess symptoms experienced in the 2 weeks prior to assessment, such as intense sadness, crying, or changes in sleep, appetite, or sexual interest. Items are on a 4-point scale ranging from 0 to 3, with a maximum score of 63. Higher total scores indicate more severe depression symptoms. Administration of the scale takes about 10 minutes.
Mongomery Asberg Depression Rating Scale | 1 Day
  is a 10-items questionnaire that is used to measure the core symptoms and cognitive features of clinical depression (33). An higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. The subject has to be interviewed by a trained psychologist or psychiatrist.
Symbol Digit Modalities Test | 1 Day
  is a measure of attention and processing speed. It presents a series of nine symbols, each of which is paired with a single digit, labelled 1-9, in a key at the top of a sheet. The remainder of the page has a pseudorandomized sequence of the symbols and the subject must respond with the digit associated with each of these as quickly as possible. The score is the number of correct answers in 90 seconds.
Paced Auditory Serial Addition Test | 1 Day
  is another measure of sustained attention and speed of information processing. The subject hears a series of single digit number from CD that are presented at the rate of one every 3 seconds in the first part of the test (PASAT 3"), or at the rate of one every 2 seconds in the second part (PASAT 2"). The subject is asked to add each consecutive digit to the one immediately preceding it. Sixty-one digits are presented for each part and each part has a maximum of 60 correct answers.
Stroop Test | 1 Day
  evaluates sustained attention and some aspects of executive functions, such as the ability to elaborate relevant and irrelevant dimensions in parallel and to inhibit an automatic response while performing a task based on conflicting stimuli. The procedure comprised of three trials. In the first trial, the subject is instructed to read a list of word indicating colours printed in black ink as quickly as possible; in the second trial the subject is instructed to name the colour of strings of dots as quickly as possible; in the third trial (interference condition), the subject has to name the colours of the ink of words indicating conflicting colours as quickly as possible. Performance will assess by calculating the time required to name the items and the number of the errors.

OTHER OUTCOMES:
State-Trait Anxiety Inventory Form Y | 1 Day
  is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndrome. Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale. Higher scores indicate greater anxiety. Administration of the questionnaire take about 10 minutes.
SCID-I Disorders- Patient Edition | 1 Day
  semi-structured interview for making the major DSM-IV Axis I diagnoses. It contains the following modules: Mood Episodes, Psychotic and Associated Symptoms, Psychotic Disorders, Mood Disorders, Substance Use Disorders, Anxiety Disorders, Somatoform Disorders, Eating Disorders, and Adjustment Disorder. Each criterion is coded as either ?,1,2, or 3 (?= inadequate information to code the criterion; 1= the symptom described in the criterion is clearly absent; 2= the threshold for the criterion is almost, but not quite, met; 3= the threshold for the criterion is just met.).
Selective Reminding Test | 1 Day
  assess verbal learning and delayed recall. It include a list of 12 words and uses six consecutive learning trials and a delayed trials A word recalled on two consecutive trials is considered to have a long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total sum of the words in LTS of all six trials is taken (SRT-LTS). If a word in LTS is consistently recalled on all subsequent trials, it is then scored as in Consistent Long Term Retrieval (CLTR). The total sum of the word in CLTR of all six trials is taken (SRT-CLTR). The Delayed Recall (SRT-D) is the total number of words recalled after the delayed period.
10/36 Spatial Recall Test | 1 Day
  assess visuo-spatial learning and delayed recall. In the test, a checkerboard, with ten checkers arranged in a particular pattern, is shown to the subject for ten second. Then the subject is asked to reproduce the same pattern with ten checkers on an empty checkerboard. The test includes three consecutive trials and a delayed trials. The score is the number of correct responses for the three trials and a delayed recall trials (SPART-D).
Word List Generation | 1 Day
  explores verbal fluency on semantic stimulus by asking the subject to produce as many words as possible belonging to a semantic category within 90 seconds. The score is the number of correct words.
Pittsburgh Sleep Quality Index | 1 Day
  a self-rated questionnaire which differentiates "poor" from "good" sleepers by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction (27). Scoring of the answers is based on a 0 to 3 scale, where 3 reflects the negative extreme on the Likert Scale. The sum of the seven sub-scores generates the total score where 5 is the cut-off for distinguishing poor (higher) from good (lower) sleepers. The PSQI has internal consistency and a reliability coefficient (Cronbach's alpha) of 0.83 for its seven components.
Psychomotor Vigilance Task | 1 Day
  it is a sustained-attention, reaction-timed task that is easily used to test the speed with which subjects respond to a visual stimulus, by pressing a button (28). It has become a standard laboratory tool in a variety of experimental conditions and in the sleep lab it is commonly used to assess the effects of sleep restriction on sustained performance (29-31). The PVT is a simple task where the subject is placed in front of a monitor where a light randomly appears every few seconds for 10 minutes and is asked to press a button as soon as the light appears. The main measurement is to see how many times the button is not pressed when the light is on. The test gives a numerical measure of sleepiness by counting the number of lapses in attention.
Multiple Sclerosis quality of life (MSQol-54) | 1 Day
  it is one of the most widely used MS-specific health related quality of life, instruments (34). This questionnaire includes 54 items distributed into multi-item scales (Physical health, Physical role limitations, Emotional role limitations, Pain, Emotional well-being, Energy, Social function, Cognitive function, Health perception, Health distress, Overall quality of life, Sexual function) and two single items (Change in health, Sexual function satisfaction). Two summary scores-physical health composite and mental health composite can be derived from a weighted combination of scale scores. MSQol-54 scale scores will create using the Likert method by averaging items within the scales, and then row scores will be linearly transformed into 0-100 scales. Higher values indicate better quality of life.
Sleep parameter time in bed | 1 Day
Sleep parameter Total Sleep Time (min) | 1 Day
Sleep parameter Sleep efficiency (% TST/Time spent in bed) | 1 Day
Sleep parameter Wake after sleep onset | 1 Day
Sleep parameter Number of awakenings | 1 Day
Sleep parameter Stage N1 (% of TST) | 1 Day
Sleep parameter Stage N2 (% of TST) | 1 Day
Sleep parameter Stage N3 (% of TST) | 1 Day
Sleep parameter Stage REM (% of TST) | 1 Day
Sleep parameter Total arousal index | 1 Day
Sleep parameter Limb movements index (nr/hour of sleep) | 1 Day
Sleep parameter Periodic limb movement index (nr/hr of sleep) | 1 Day
Sleep parameter Apnea/hypopnea Index (nr/hr of sleep) | 1 Day
Sleep parameter Oxygen desaturation index (nr of desaturations ≥ 4% /hr of sleep) | 1 Day
Sleep parameter Cyclic alternating pattern rate | 1 Day
Sleep parameter Phases A1 rate (nr/hr of non-REM) | 1 Day
Sleep parameter Phases A2 rate (nr/hr of non-REM) | 1 Day
Sleep parameter Phases A3 (nr/hr of non-REM) | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Gobbi, MD, Principal Investigator — Ospedale Regionale di Lugano - Civico
Locations (1):
- Ospedale Regionale di Lugano - Civico, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kos D, Kerckhofs E, Nagels G, D'hooghe MB, Ilsbroukx S. Origin of fatigue in multiple sclerosis: review of the literature. Neurorehabil Neural Repair. 2008 Jan-Feb;22(1):91-100. doi: 10.1177/1545968306298934. Epub 2007 Apr 4. PMID 17409388
- [Background] Bamer AM, Johnson KL, Amtmann D, Kraft GH. Prevalence of sleep problems in individuals with multiple sclerosis. Mult Scler. 2008 Sep;14(8):1127-30. doi: 10.1177/1352458508092807. Epub 2008 Jul 16. PMID 18632776
- [Background] Attarian HP, Brown KM, Duntley SP, Carter JD, Cross AH. The relationship of sleep disturbances and fatigue in multiple sclerosis. Arch Neurol. 2004 Apr;61(4):525-8. doi: 10.1001/archneur.61.4.525. PMID 15096400
- [Background] Mohr DC, Hart SL, Goldberg A. Effects of treatment for depression on fatigue in multiple sclerosis. Psychosom Med. 2003 Jul-Aug;65(4):542-7. doi: 10.1097/01.psy.0000074757.11682.96. PMID 12883103
- [Background] Jongen PJ, Ter Horst AT, Brands AM. Cognitive impairment in multiple sclerosis. Minerva Med. 2012 Apr;103(2):73-96. PMID 22513513
- See also: Official website of facility — http://www.eoc.ch
- See also: Official website of funding organisation — https://www.multiplesklerose.ch/